CLINICAL TRIAL: NCT05943132
Title: MISC-CBO: a Cluster Randomized Control Trial to Improve the Mental Health of OVC in South Africa
Brief Title: MISC-CBO to Improve the Mental Health of OVC in South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Carla Sharp, Director of the Developmental Psychopathology Lab Clinical Psychology, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003813
Record Dates: First submitted 2023-06-22; First posted 2023-07-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Mental Disorder, Child
Keywords: mental health problems; Mediational Intervention for Sensitizing Caregivers; mentalizing; caregivers
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 24 Community-based Organizations (CBOs) (360 children), their caregivers at home and 72 CBO caseworkers are enrolled. Randomization takes place at the level of the CBO so that half of the CBOs receive MISC and the other half receives TAU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MISC-CBO (Experimental): MISC-CBO is a year-long semi-structured, manualized video-feedback caregiver intervention that targets key components in caregiver-child interactions known to improve caregiving quality and child outcomes. These components include emotional and cognitive components shown to improve socio-emotional and cognitive developmental outcomes in children.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC)
- Treatment as Usual (Other): TAU at CBOs include provision of meals, counselling services mostly focused on social support, financial assistance, and healthcare counseling - all which promote the mental health of OVC, but does not include a specific focus on caregiving quality.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC) — MISC-CBO is a year-long semi-structured, manualized video-feedback caregiver intervention that targets key components in caregiver-child interactions known to improve caregiving quality and child outcomes. These components include emotional and cognitive components shown to improve socio-emotional and cognitive developmental outcomes in children.
  Other Names: mentalization-based intervention
  Arms: MISC-CBO
Behavioral: Treatment as Usual — Treatment as Usual includes general support for children in homework and nutrition.
  Arms: Treatment as Usual

SUMMARY:
The goal of this cluster randomized control clinical trial is to evaluate the effectiveness of the Mediational Intervention for Sensitizing Caregivers for Community-based Organizations (MISC-CBO) in reducing mental health problems in orphan and vulnerable children in South Africa.

Aim 1 will evaluate the direct effects of MISC-CBO on video-coded CBO caseworker caregiving quality (affiliation and attachment) and children's mental health outcomes over a 24 month period. 24 CBOs (360 children and 72 caseworkers) will be recruited using existing Non-Governmental Organization (NGO) partner (Childline) in two districts in the Free State, South Africa (SA). CBOs will be randomly assigned to receive either one year of bi-weekly MISC-CBO or Treatment as Usual (TAU). The investigators hypothesize that MISC-CBO will be associated with comparative increases in caseworker caregiving quality and reductions in mental health problems in Orphans and Vulnerable Children (OVC).

Aim 2a,will test the hypothesis that caregiving quality at end-of-intervention (12 months) accounts for intervention effects on child mental health at 18 and 24 months. Aim 2b will evaluate the moderating effects of orphan status and the quality of the home environment, expecting that OVC who are maternal and double orphans, and from impoverished home environments will show reduced response to intervention compared to children without these risk factors.

Aim 3a will use World Health Organization metrics to test the hypothesis that MISC-CBO is cost-effective in terms of disability-adjusted life years (DALYs) averted. Aim 3b will use qualitative methodology to test the hypothesis that community stakeholders deem the climate favorable and ready for the implementation of MISC-CBO, and that additional barriers and facilitators for scale-up and implementation will be identified.

The proposed work extends the investigators' formative work to now fully test the real-world effectiveness, mechanisms of action, cost-effectiveness and implementation readiness of MISC-CBO during the critical developmental window of at-risk children aging into adolescence, consistent with National Institute of Mental Health's strategic objectives.

DETAILED DESCRIPTION:
The negative impact of acquired immunodeficiency syndrome (HIV/AIDS) on child mental health through orphanhood, parental chronic illness and poverty is well documented. These interconnecting factors led to the operational term "orphans and vulnerable children" (OVC). Currently, there are +16 million OVC, the vast majority in sub-Saharan Africa (SSA), with estimates between 1.95-3.7 million in South Africa (SA). Given the scarcity of mental health workers in SSA, community-based organizations (CBOs) offer a strategic point of intervention as an essential response to shortages in human resources for mental health. However, as yet, no Randomized Control Trial (RCT) has evaluated the effects of improving the quality of caregiving of CBO caseworkers in their daily interactions with children, conferring a missed opportunity to leverage the CBO environment directly to improve child mental health. Over the past 5 years, the investigators have successfully adapted and implemented the Mediational Intervention for Sensitizing Caregivers for CBOs building on Co-Investigator Boivin's parent-based RCTs in Uganda . MISC adapted for CBOs (MISC-CBO) is a year-long semi-structured, manualized video-feedback intervention designed to enhance the caregiving capacity of CBO caseworkers to improve child outcomes, by targeting the Research Domain Criteria systems for social processes (affiliation and attachment) in daily caseworker-child interactions. The investigators showed that MISC-CBO significantly improved caregiving quality and mental health outcomes of OVC over a 12-month period12. However, the study was a quasi-experimental feasibility trial that limits causal conclusions, did not have statistical power to detect mediating and moderating effects, did not follow up with children beyond post-intervention, and did not assess cost-effectiveness or implementation climate and readiness. Consistent with the Research Domain Criteria's dimensional approach to psychopathology, the overall goal of the proposed study is to conduct a repeated measures cluster randomized control trial to fully establish the effectiveness and trans-diagnostic mechanisms of action of MISC-CBO in high risk 7-11 year olds - a developmental stage critical for building mental health resilience against the adolescent onset of psychiatric problems. 24 CBOs will participate, each with 15 OVC and 3 caseworkers, recruited using existing NGO partner (Childline) and infrastructure in two districts in the Free State, SA, totaling 360 children (50% female; 7-11 year old, equal age bands) and 72 CBO caseworkers (100% female). The 24 CBOs will be randomly assigned to receive either one year of bi-weekly MISC-CBO or TAU. Video-based observations of caseworker caregiving quality and multi-informant child mental health will be assessed at baseline, 12 (end-of-intervention time point), 18 and 24 months. Next, the investigators will use Consolidated Framework for Implementation Research (CFIR13) constructs and input from a Community Advisory Board (CAB) to leverage the RCT to evaluate implementation costs, climate and readiness that would better position the RCT results for future uptake, scale up, and sustainability.

Aim 1. Evaluate the direct effects of MISC-CBO on child mental health. Hypotheses include that CBO caseworkers assigned to MISC-CBO vs. TAU will show continued improvement in quality of caregiving at post-intervention (12 months), 18 months, and 24 months follow-up and that children assigned to MISC-CBO vs. TAU will show continued and significant reductions in mental health symptoms at 12 months, 18 months, and 24 months follow-up.

Aim 2. Evaluate improved caregiving as mediator of follow-up outcomes (Aim 2a) and child and home characteristics as moderators of MISC-CBO vs. TAU intervention effects (Aim 2b). The investigators hypothesize that reduction in child mental health symptoms at 18 and 24 months will be mediated by improved CBO caseworker caregiving quality observed through video at post intervention (12 months), and that positive effects of MISC-CBO vs. TAU at 12, 18 and 24 months will be reduced for maternal and double orphans, and children from impoverished home environments compared to children without these risk characteristics.

Aim 3. Evaluate the cost-effectiveness of MISC-CBO for improved child mental health (Aim 3a) and evaluate implementation climate and readiness for future scale-up (Aim 3b). For Aim 3a, the investigators will follow World Health Organization (WHO) metrics to determine the cost-effectiveness of public health interventions through assessment of disability-adjusted life years (DALYs) averted. The investigators hypothesize that MISC-CBO will prove a cost-effective method to improve child mental health. For Aim 3b, the investigators will conduct three focus groups (each n=7 to total 21) with representatives from the government sector (Departments of the Free State Provincial Government), non-governmental or organized civil society (Non-Governmental Organizations and CBOs) and the University sector (Departments of Psychology and Education), at post-intervention (12 months post baseline). The investigators hypothesize that relevant community stakeholders will deem the climate favorable and ready for the implementation and scale-up of MISC-CBO, and that additional barriers and facilitators for scale-up and implementation will be identified.

Study impact. The proposed work will test the real-world effectiveness, mechanisms of action, cost-effectiveness and implementation readiness of a culturally sensitive, community-based mental health intervention, MISC-CBO, during the critical developmental window of at-risk children aging into adolescence. The program of research is therefore in line with the third strategic objective of the National Institute of Mental Health ("Strive for prevention and cure") that articulates the need for validated targets for interventions, and improved methods to match interventions to under-served individuals and populations that can be scaled for greater public health impact.

ELIGIBILITY:
Inclusion Criteria:

1. Status as OVC.
2. Children will be 7-11 years old
3. Resident in the CBO catchment area
4. Child has a legal guardian

Exclusion Criteria:

1. Children with a medical history of serious birth complications
2. Children with a medical history severe malnutrition
3. Children with a neurological disability

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 792 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Mental health problems | Repeated measures: baseline, and again 12, 18, 24 months post baseline
  Reduced mental health problems in children will be assessed by the Strengths and Difficulties Questionnaire (SDQ). The is a multi-informant 25-item measure of emotional and behavioral disorders for children aged 3-17 widely used across the world. Both informant and youth versions of the SDQ utilize a three-point Likert scale ranging from 'not true (0)', 'somewhat true' (1), to 'certainly true' (2). The use of a total difficulties score is common as a general index of mental health problems. Scores may range from 0 to 60 with higher scores indicating increased mental health problems.
Quality of caregiving capacity in CBO caseworkers | Repeated measures: baseline, and again 12 (end-of-intervention), 18 and 24 months post baseline
  Improved quality caregiving is measured by a standardized MISC videotaped observational tool, the Observing Mediational Interaction (OMI). The OMI is an observational tool that counts the number of times caregivers engage in behaviors that promote cognitive and social development in children. As such, it has a minimum range of 0; however it has no upper range as any number of behaviors may be coded during an interaction. Increased frequency of sensitive behaviors indicates increased quality of caregiving.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Free State, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: Undecided